CLINICAL TRIAL: NCT03174184
Title: A Phase 2a Study of the Early Bactericidal Activity of Rifampin (RIF) in Combination With Meropenem Plus Amoxicillin/Clavulanate Among Adults With Rifampin-resistant or Rifampin-susceptible Pulmonary Tuberculosis
Brief Title: Early Bactericidal Activity of Rifampin + Meropenem + Amoxicillin/Clavulanate in Adults With Pulmonary TB
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB00119017; FD-R-05724 (Other Grant/Funding Number: FDA OOPD)
Record Dates: First submitted 2017-05-30; First posted 2017-06-02 (Actual); Results first posted 2023-07-19 (Actual); Last update posted 2023-07-19 (Actual); Status verified 2023-06

CONDITIONS: Tuberculosis, Pulmonary
MeSH Terms: conditions — Tuberculosis, Pulmonary | interventions — Rifampin; Rifamycins; Meropenem; Amoxicillin; Clavulanic Acid; Amoxicillin-Potassium Clavulanate Combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- Rifampin resistant A (Experimental): Participants with the presence of rifampin resistance-conferring rpoB mutations in M. tuberculosis who will receive RIFAMPIN 20mg/kg once daily (QD), MEROPENEM 2 grams (G) thrice daily (TID) intravenously, Amoxicillin/Clavulanate Potassium 500 milligrams (MG)-125 MG Oral Tablet once daily for 14 days
  Interventions: Drug: Rifampin; Drug: MEROPENEM 2 grams TID; Drug: Amoxicillin/Clavulanate Potassium 500 MG-125 MG Oral Tablet
- Rifampin resistant B (Experimental): Participants with the presence of rifampin resistance-conferring rpoB mutations in M. tuberculosis who will receive MEROPENEM 2 grams TID (thrice daily) intravenously, Amoxicillin/Clavulanate Potassium 500 MG-125 MG Oral Tablet once daily for 14 days
  Interventions: Drug: MEROPENEM 2 grams TID; Drug: Amoxicillin/Clavulanate Potassium 500 MG-125 MG Oral Tablet
- Rifampin susceptible C (Experimental): Participants without the presence of rifampin resistance-conferring rpoB mutations in M. tuberculosis who will receive RIFAMPIN 20mg/kg once daily, MEROPENEM 2 grams TID (thrice daily) intravenously, Amx/Clv orally at a dose of 500 mg/125 mg thrice daily for 14 days
  Interventions: Drug: Rifampin; Drug: MEROPENEM 2 grams TID; Drug: Amoxicillin/Clavulanate Potassium 500 MG-125 MG Oral Tablet
- Rifampin susceptible D (Experimental): Participants without the presence of rifampin resistance-conferring rpoB mutations in M. tuberculosis who will receive MEROPENEM 2 grams TID intravenously, Amoxicillin/Clavulanate Potassium 500 MG-125 MG Oral Tablet once daily for 14 days
  Interventions: Drug: MEROPENEM 2 grams TID; Drug: Amoxicillin/Clavulanate Potassium 500 MG-125 MG Oral Tablet
- Rifampin susceptible E (Experimental): Participants without the presence of rifampin resistance-conferring rpoB mutations in M. tuberculosis who will receive MEROPENEM 1 gram TID intravenously, Amoxicillin/Clavulanate Potassium 500 MG-125 MG Oral Tablet once daily for 14 days
  Interventions: Drug: MEROPENEM 1 gram TID; Drug: Amoxicillin/Clavulanate Potassium 500 MG-125 MG Oral Tablet
- Rifampin susceptible F (Experimental): Participants without the presence of rifampin resistance-conferring rpoB mutations in M. tuberculosis who will receive MEROPENEM 3 grams QD intravenously, Amoxicillin/Clavulanate Potassium 875 MG-125 MG Oral Tablet once daily for 14 days
  Interventions: Drug: MEROPENEM 3 grams QD; Drug: Amoxicillin/Clavulanate Potassium 875 MG-125 MG Oral Tablet

INTERVENTIONS:
Drug: Rifampin — Oral administration of rifampin at a dosage of 20 mg/kg daily
  Other Names: Rifamycins
  Arms: Rifampin resistant A; Rifampin susceptible C
Drug: MEROPENEM 2 grams TID — Intravenous administration at a dosage of 2 grams thrice daily
  Other Names: Merrem
  Arms: Rifampin resistant A; Rifampin resistant B; Rifampin susceptible C; Rifampin susceptible D
Drug: MEROPENEM 1 gram TID — Intravenous administration at a dosage of 1 gram thrice daily
  Other Names: Merrem
  Arms: Rifampin susceptible E
Drug: MEROPENEM 3 grams QD — Intravenous administration at a dosage of 3 grams once daily
  Other Names: Merrem
  Arms: Rifampin susceptible F
Drug: Amoxicillin/Clavulanate Potassium 500 MG-125 MG Oral Tablet — Amx/Clv will be administered orally at a dose of 500 mg/125 mg thrice daily
  Other Names: Augmentin
  Arms: Rifampin resistant A; Rifampin resistant B; Rifampin susceptible C; Rifampin susceptible D; Rifampin susceptible E
Drug: Amoxicillin/Clavulanate Potassium 875 MG-125 MG Oral Tablet — Amx/Clv will be administered orally at a dose of 875 mg/125 mg once daily
  Other Names: Augmentin
  Arms: Rifampin susceptible F

SUMMARY:
The overall goal of this exploratory proof-of-concept study is to determine whether, in participants with pulmonary tuberculosis caused by M. tuberculosis (MTB) with or without rifampin resistance-conferring rpoB-gene mutations, the combination of meropenem and amoxicillin/clavulanate with rifampin has greater early bactericidal activity (EBA) than the combination of meropenem and amoxicillin/clavulanate without rifampin. Funding Source- FDA OOPD.

DETAILED DESCRIPTION:
This is a proof-of-concept study to determine whether, in humans infected with M. tuberculosis that is resistant or susceptible to rifampin based on conventional drug susceptibility testing, the combination of meropenem, amoxicillin/clavulanate, and rifampin has activity that is sufficiently promising to proceed with further drug development along these lines. Rifampin has an incompletely understood but critical role in eradication of M. tuberculosis persisters and consequently the shortening of the duration of treatment for 'rifampin susceptible' tuberculosis (TB). For Multi-Drug Resistant (MDR) / Extensively Drug Tuberculosis (XDR) TB, the ability to recoup rifampin's antituberculosis activity through rational combination with a carbapenem and a β-lactamase inhibitor with or without amoxicillin could transform the treatment of this disease.

This proof-of-concept study is designed such that a negative outcome would refute the hypothesis that the combination of a carbapenem and amoxicillin/clavulanate with rifampin will have greater activity than either component alone against M. tuberculosis strains having Minimum Inhibitory Concentrations (MIC) in the range considered resistant to rifampin. A positive study outcome would catalyze further research to identify optimal dosing strategies for all regimen components as well as development of carbapenems optimized for TB treatment with respect to targets of activity, stability against hydrolysis, and oral formulation.

The study hypothesis cannot be tested satisfactorily in traditional animal models of tuberculosis chemotherapy due to the rapid inactivation of carbapenems (as well as other beta-lactams) by dehydropeptidases that are expressed at high levels in mouse, rabbit, and guinea pig tissues. However, all of the study drugs are Food and Drug Administration (FDA) -approved for various infectious disease indications, are in routine clinical use, and have good safety profiles, such that proceeding with the proposed clinical trial based on in vitro data is justified.

This study will also characterize the relationship between meropenem exposure (in combination with amoxicillin/clavulanate) and early bactericidal activity in order to identify the pharmacokinetic drivers of activity and pharmacokinetic targets for desired effects. This will inform the identification of more feasible meropenem dosing strategies in the near term, as well as the dose selection for novel oral carbapenems that may be available for tuberculosis treatment in the future. The proportion of the dosing interval for which free drug concentrations exceed MIC (T>MIC) is the pharmacokinetic (PK) / pharmacodynamic(PD) parameter most closely correlated with efficacy of carbapenems against common fast-growing bacteria such as Enterobacteriaceae that cause infections for which meropenem is currently approved. A commonly accepted target for efficacy in these infections is 40% T>MIC, which requires multiple daily doses to achieve. Whether this PK/PD parameter and target value is optimal for carbapenem treatment of infections with M. tuberculosis, which has a much longer doubling time, is unknown. In the trial by Diacon et al, meropenem 2 grams thrice daily plus amoxicillin/clavulanate resulted in a median T>MIC of 76% [90% Confidence Interval (CI): 66-93] whereas faropenem sodium 600 mg thrice daily plus amoxicillin/clavulanate resulted in T>MIC of 13% (90% CI: 0-33), indicating that if T>MIC is the single parameter most strongly linked to efficacy in tuberculosis, then the target for bactericidal effect is between 13% and 76%, and lower and/or less frequent doses (or use of oral carbapenems with lower bioavailability) may still have significant efficacy. If T>MIC is not the efficacy-linked PK/PD parameter, less frequent administration of the same total dose is likely to remain equally effective.

ELIGIBILITY:
Inclusion Criteria:

* New or recurrent pulmonary TB with one or both of the following:
* sputum positive for acid-fast bacilli on direct microscopy of at least grade 1+ (International Union Against Tuberculosis and Lung Disease (IUATLD) scale) on at least one pre-treatment sputum sample
* sputum positive for M. tuberculosis by Xpert® MTB/RIF testing, with semiquantitative result of 'medium' or 'high' on at least one pre-treatment sputum sample
* Age ≥18 and ≤65 years at study screening
* Ability and willingness to provide informed consent
* Body weight 40 kg to 90 kg, inclusive
* Laboratory values obtained within 30 days prior to or at study screening:
* Absolute neutrophil count (ANC) > 750 cells/mm3
* Hemoglobin 7.0 g/dL
* Platelet count 50,000/mm3
* Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤ 3 X upper limit of normal (ULN)
* Total bilirubin ≤ 2.5 X ULN
* Creatinine < 1.5 X ULN
* HIV infection must be documented as either absent or present
* For HIV-positive candidates only: CD4+ cell count of ≥ 100 cells/cu mm, performed within 30 days prior to or at study screening
* For females of reproductive potential, negative serum or urine pregnancy test within 7 days prior to or at study screening. Female participants who are participating in sexual activity that could lead to pregnancy must agree to use one reliable non-hormonal method of contraception (condoms or an IUD), or another method (diaphragm or cervical cap) if it is approved by the national regulatory authority and used according to package insert, while receiving study medications.
* Willingness to be hospitalized for a minimum of 16 consecutive days
* Ability to produce an overnight sputum sample of sufficient quality and quantity. As a guideline, this should be 10 ml or more during a 16-hour collection period. Volume is clinically estimated from a spot sample provided at screening and verified upon the first overnight collection (which can be repeated upon retraining).
* Xpert® MTB/RIF result performed on sputum within 14 days prior to or at study screening that shows EITHER 'Rifampin resistance detected' OR 'Rifampin resistance not detected'

Exclusion Criteria:

* Treatment with any drug active against M. tuberculosis within the 3 months prior to study screening.
* Breast-feeding
* Known allergy or sensitivity to any of the study drugs
* Participants receiving valproate sodium or probenecid
* Karnofsky score < 60 OR poor general condition such that, in the opinion of the investigator at screening, any delay in initiation of definitive TB treatment cannot be tolerated
* Known current neurological TB or seizure disorder
* Any condition as determined by physical examination, medical history, laboratory data, or chest x-ray which, in the opinion of the investigator, would interfere with safety or endpoint assessments in the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 112 (Actual)
Dates: Start 2017-08-23 (Actual); Primary Completion 2022-05-13 (Actual); Study Completion 2022-05-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kelly Dooley, MD, Principal Investigator — Associate Professor of Medicine
Locations (1):
- Task Applied Science and Stellenbosch University, Stellenbosch, South Africa

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] De Jager V, Gupte N, Nunes S, Barnes GL, van Wijk RC, Mostert J, Dorman SE, Abulfathi AA, Upton CM, Faraj A, Nuermberger EL, Lamichhane G, Svensson EM, Simonsson USH, Diacon AH, Dooley KE. Early Bactericidal Activity of Meropenem plus Clavulanate (with or without Rifampin) for Tuberculosis: The COMRADE Randomized, Phase 2A Clinical Trial. Am J Respir Crit Care Med. 2022 May 15;205(10):1228-1235. doi: 10.1164/rccm.202108-1976OC. PMID 35258443

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Rifampin Resistant A | Rifampin Resistant B | Rifampin Susceptible C | Rifampin Susceptible D | Rifampin Susceptible E | Rifampin Susceptible F
Started | 32 | 20 | 17 | 15 | 14 | 14
Completed | 23 | 15 | 12 | 12 | 12 | 12
Not Completed | 9 | 5 | 5 | 3 | 2 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Rifampin Resistant A | Rifampin Resistant B | Rifampin Susceptible C | Rifampin Susceptible D | Rifampin Susceptible E | Rifampin Susceptible F | Total
Number analyzed (Participants) | 32 | 20 | 17 | 15 | 14 | 14 | 112
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 37 [27 to 44] | 37 [30 to 47] | 33 [26 to 47] | 36 [33 to 45] | 45 [30 to 47] | 34 [30 to 43] | 36 [28 to 46]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 5 | 4 | 7 | 2 | 2 | 32
  Male | 20 | 15 | 13 | 8 | 12 | 12 | 80
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 13 | 9 | 3 | 2 | 5 | 7 | 39
  White | 0 | 0 | 0 | 0 | 0 | 0 | 0
  More than one race | 19 | 11 | 14 | 13 | 9 | 7 | 73
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  South Africa | 32 | 20 | 17 | 15 | 14 | 14 | 112
HIV positive [Count of Participants; unit: Participants] | 9 | 5 | 2 | 4 | 3 | 6 | 29
BMI [Median (Inter-Quartile Range); unit: kg/m^2] | 18.3 [17.5 to 20.0] | 17.8 [16.6 to 19.9] | 18.9 [17.9 to 20.1] | 18.7 [17.1 to 19.7] | 19.4 [18.2 to 20.8] | 18.1 [16.6 to 19.8] | 18.4 [17.3 to 20.2]
MGIT Time to Positivity [Median (Inter-Quartile Range); unit: Days] | 4.8 [3.9 to 6.3] | 5.8 [4.1 to 7.7] | 4.3 [3.8 to 7.4] | 4.4 [3.8 to 5.7] | 5.7 [4.3 to 6.4] | 4.9 [3.9 to 7.3] | 4.8 [3.9 to 6.6]

OUTCOME MEASURES:

1. Primary Outcome: Estimate of the 14-day Early Bactericidal Activity (EBA), Based on Colony Forming Unit Counts, of the Combination of Meropenem and Amoxicillin/Clavulanate, Without Versus With Rifampin
Description: The Early Bactericidal Activity (EBA) over a 14 days period (EBA0-14), as determined by the median rate of change in log10 Colony Forming Units (CFU) per mL sputum. A non-linear mixed effects model of log10 CFU/mL sputum on time was developed using aggregated participant data for each treatment arm. A basic model was developed based on mono- or bi-exponential bacterial killing functions. Afterwards, covariate modelling to identify relationships between demographics, disease severity, secondary pharmacokinetic summary indices (area under the curve from time 0 to last measured concentration (AUC0-last) and maximum observed plasma concentration (Cmax), and model parameters describing log10 CFU/mL sputum over time was performed. Finally, the treatment regimen was tested using different functions supported by the graphical analysis.
Time Frame: 14 days
Population: EBA could not be calculated among some participants who did not complete dosing
Measure: Mean (95% Confidence Interval); unit: rate of change in log10 CFU/mL/day
Arm/Group | Rifampin Resistant A | Rifampin Resistant B | Rifampin Susceptible C | Rifampin Susceptible D | Rifampin Susceptible E | Rifampin Susceptible F
Number analyzed (Participants) | 22 | 17 | 14 | 15 | 12 | 14
rate of change in log10 CFU/mL/day | -0.06 [-0.09 to -0.02] | -0.11 [-0.15 to -0.0] | -0.14 [-0.20 to -0.08] | -0.12 [-0.16 to -0.08] | -0.05 [-0.09 to -0.004] | -0.02 [-0.06 to 0.03]
Statistical Analysis 1: Comparison: Rifampin Resistant A vs Rifampin Resistant B vs Rifampin Susceptible C vs Rifampin Susceptible D vs Rifampin Susceptible E vs Rifampin Susceptible F; Test type: Equivalence — Equivalence tests will be conducted to examine whether the EBA0-14CFU of Arm A is different from the EBA0-14CFU of Arm B. A similar comparison will be done comparing Arm C to Arm D, Arm A to Arm C, Arm D to Arm E, Arm D to Arm F, and Arm E to Arm F; p < 0.001, Regression, Linear

2. Primary Outcome: AUC for Rifampin
Description: Rifampin AUC0-last in Arms A and C
Time Frame: 14 days
Population: Participants in Arms B, D, E, and F did not receive rifampicin. In Arm A, some participants dropped out prior to PK collection day
Measure: Mean (Full Range); unit: h*mg/L
Arm/Group | Rifampin Resistant A | Rifampin Resistant B | Rifampin Susceptible C | Rifampin Susceptible D | Rifampin Susceptible E | Rifampin Susceptible F
Number analyzed (Participants) | 23 | 0 | 12 | 0 | 0 | 0
h*mg/L | 105 [52 to 226] |  | 109 [82 to 136] |  |  |

3. Secondary Outcome: Frequency of Grade 2 or Higher Adverse Events
Description: Grade 2 or higher Adverse Events (AE) that constitute any untoward medical occurrence in a study participant and which does not necessarily have a causal relationship with this treatment. An adverse event can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of a medicinal product, whether or not related to the medicinal product.
Time Frame: From the time a study participant receives the first dose of study drug through the final study visit, up to 28 days
Measure: Number; unit: Events
Arm/Group | Rifampin Resistant A | Rifampin Resistant B | Rifampin Susceptible C | Rifampin Susceptible D | Rifampin Susceptible E | Rifampin Susceptible F
Number analyzed (Participants) | 32 | 20 | 17 | 15 | 14 | 14
Events | 28 | 15 | 5 | 8 | 3 | 7

4. Secondary Outcome: Distribution of Minimum Inhibitory Concentration (MIC) of Rifampin
Description: The distribution of rifampin MIC in the drug-resistant arms
Time Frame: 14 days
Population: Rifampin MIC was only measured in Arms A and B. Some cultures did not grow in subculture and MIC could not be assessed in Arms A and B.
Measure: Median (Full Range); unit: mcg/mL
Arm/Group | Rifampin Resistant A | Rifampin Resistant B | Rifampin Susceptible C | Rifampin Susceptible D | Rifampin Susceptible E | Rifampin Susceptible F
Number analyzed (Participants) | 30 | 16 | 0 | 0 | 0 | 0
mcg/mL | 1.28 [0.32 to 1.28] | 1.28 [0.32 to 1.28] |  |  |  |

5. Secondary Outcome: Estimate the Antimycobacterial Activity Based on Liquid Culture Time-to-positivity
Description: Change in time-to-positivity in Mycobacteria Growth Indicator Tube (MGIT) liquid media over 14 days of treatment (EBA0-14(TTP)) (time to positivity) for the study treatments. The Early Bactericidal Activity (EBA) over a 14 days period (EBA0-14), as determined by the median rate of change in TTP (expressed in log10 hours/day). A non-linear mixed effects model of log10 hours/day on time was developed using aggregated participant data for each treatment arm. A basic model was developed based on mono- or bi-exponential bacterial killing functions. Afterwards, covariate modelling to identify relationships between demographics, disease severity, secondary pharmacokinetic summary indices (area under the curve from time 0 to last measured concentration (AUC0-last) and maximum observed plasma concentration (Cmax), and model parameters describing TTP over time was performed. Finally, the treatment regimen was tested using different functions supported by the graphical analysis.
Time Frame: 14 days
Population: Some participants dropped out and did not contribute enough longitudinal TTP data to contribute to these assessments
Measure: Mean (95% Confidence Interval); unit: rate of change in log10 hours/day
Arm/Group | Rifampin Resistant A | Rifampin Resistant B | Rifampin Susceptible C | Rifampin Susceptible D | Rifampin Susceptible E | Rifampin Susceptible F
Number analyzed (Participants) | 30 | 18 | 15 | 15 | 13 | 14
rate of change in log10 hours/day | 0.19 [0.08 to 0.29] | 0.31 [0.19 to 0.43] | 0.53 [0.38 to 0.68] | 0.20 [0.13 to 0.27] | 0.09 [0.03 to 0.15] | 0.09 [-0.03 to 0.21]

ADVERSE EVENTS:
Time Frame: 28 days
Description: Standard AE and SAE definitions apply
Arm/Group | Rifampin Resistant A | Rifampin Resistant B | Rifampin Susceptible C | Rifampin Susceptible D | Rifampin Susceptible E | Rifampin Susceptible F
All-Cause Mortality (participants affected / at risk) | 0/32 | 0/20 | 0/17 | 0/15 | 0/14 | 0/14
Serious Adverse Events (participants affected / at risk) | 0/32 | 0/20 | 0/17 | 2/15 | 0/14 | 0/14
Other Adverse Events (participants affected / at risk) | 6/32 | 2/20 | 2/17 | 1/15 | 0/14 | 0/14
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Rifampin Resistant A (N=32) | Rifampin Resistant B (N=20) | Rifampin Susceptible C (N=17) | Rifampin Susceptible D (N=15) | Rifampin Susceptible E (N=14) | Rifampin Susceptible F (N=14)
Elevated ALT (Hepatobiliary disorders) | 0 | 0 | 0 | 1 | 0 | 0 — Grade 2 elevation of ALT and AST that led to prolongation of hospitalization
Elevated AST (Hepatobiliary disorders) | 0 | 0 | 0 | 1 | 0 | 0 — Grade 2 elevation of ALT and AST that led to prolongation of hospitalization
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Rifampin Resistant A (N=32) | Rifampin Resistant B (N=20) | Rifampin Susceptible C (N=17) | Rifampin Susceptible D (N=15) | Rifampin Susceptible E (N=14) | Rifampin Susceptible F (N=14)
Gastrointestinal side effects (Gastrointestinal disorders) | 6 | 2 | 2 | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-11-08): https://cdn.clinicaltrials.gov/large-docs/84/NCT03174184/Prot_SAP_000.pdf